CLINICAL TRIAL: NCT06136481
Title: A Pilot Randomized Control Trial of Cognitive Processing Therapy for Mental Health Problems in Earthquake Exposed Adults.
Brief Title: The Feasibility of Cognitive Process Therapy in Earthquake-affected Population With Mental Health Problems in Türkiye
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Koç University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023.240.IRB3.110
Record Dates: First submitted 2023-11-13; First posted 2023-11-18 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2024-10

CONDITIONS: Post Traumatic Stress Disorder; Depressive Symptoms; Well-Being, Psychological; Anxiety Disorders and Symptoms
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depression; Psychological Well-Being; Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Participants will not be blinded to their study arm because of the nature of the intervention, but outcome assessors will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): CPT intervention: participants will attend the 12 consecutive sessions administered by a psychologist in twice a week.
  Interventions: Other: Cognitive Processing Therapy
- Control group (No Intervention): The control (enhanced care as usual) group will receive the information about freely available psychological support options. E-CAU ranges from standard community care which may include any existing mental health support services available to earthquake survivors in container cities. The participants will be given flyers which include information about the services provided by the government and by non-governmental organizations. After completion of the post and follow-up assessment of experimental group, those in the E-CAU condition will be offered with CPT

INTERVENTIONS:
Other: Cognitive Processing Therapy — Cognitive Processing Therapy (CPT). CPT is a cognitive behavioral treatment for PTSD consisting of 12 one-hour sessions. Prior to engaging in therapy, one session will be devoted to gathering information regarding psychosocial history, trauma, and current functioning. The following sessions will follow the standard outpatient CPT protocol. The standard outpatient CPT consists of 12 one-hour sessions conducted over a 6- to 12-week period. An additional 3 weeks will be provided in case of participant and therapist vacation and/or sick days. CPT is delivered in three phases: education, processing, and challenging. The manualized treatment focuses on challenging beliefs and assumptions related to the trauma, oneself, and the world.
  Arms: Intervention group

SUMMARY:
The aim of the study is to test the pilot effectiveness of Cognitive Processing Therapy (CPT) in decreasing psychological distress and post-traumatic stress disorder (PTSD) symptoms and increasing well-being in earthquake survivors in Türkiye, using randomized controlled trial study design, which is considered the gold standard in research for evaluating the effectiveness of interventions. This pilot study will help to identify any further adaptations required prior to further effectiveness testing in a large cluster randomized controlled trial.

Study hypothesis:

Hypothesis 1: The participants who receive the CPT will have a significantly higher decrease in PTSD symptoms compared to the participants in the care-as-usual control group at the post-assessment.

Hypothesis 2: The participants who receive the CPT will have a significantly higher decrease in depressive symptom severity compared to the participants in the care-as-usual control group at the post-assessment.

Hypothesis 4: The participants who receive the CPT will have a significantly higher decrease in anxiety severity compared to the participants in the care-as-usual control group at the post-assessment.

Hypothesis 5: The participants who receive the CPT will have a significantly higher increase in well-being compared to the participants in the care-as-usual control group at post-assessment.

DETAILED DESCRIPTION:
Two large earthquakes struck Türkiye on the 6th of February 2023, affecting more than 14 million people, around 16% of the population, including more than 45.000 lost and 3.3 million displaced. Considering the current scale of the recent earthquakes in Türkiye, implementing and disseminating evidence-based psychosocial interventions, especially trauma-focused treatment approaches such as Cognitive Processing Therapy (CPT), is crucial in order to respond to the increasing mental health needs of the earthquake survivors. Cognitive Processing Therapy (CPT) is a cognitive behavioral treatment for PTSD consisting of 12 one-hour sessions. CPT is delivered in three phases: education, processing, and challenging. The manualized treatment focuses on challenging beliefs and assumptions related to the trauma, oneself, and the world. Randomized clinical trials have revealed that CPT is an effective treatment for PTSD and other comorbid conditions in a variety of civilian trauma populations.

The study will be designed as a pilot randomized controlled trial, and the potential effectiveness of individual CPT will be tested compared to the Enhanced-Care as Usual (E-CAU) control group. CPT will be implemented on Zoom, which is an online platform with HIPAA compliance. After the baseline assessment, 30 eligible participants will be randomized to two arms: in either the CPT (n =15) or only the control group (E-CAU; n=15). The first session will take place no longer than one week after the pre-intervention assessment. The post-intervention assessment through the same measures will be scheduled six weeks after the pre-intervention assessment (i.e., one week after the 12th CPT session). The follow-up assessment will be conducted one month after the post-assessment. All study participants, including dropouts, will be invited to all outcome assessments. The primary outcome is post-traumatic stress disorder, and the following are the secondary clinical outcomes: symptoms of depression, anxiety, and well-being.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or above
* Individuals who were directly impacted by earthquakes in Turkey, in February 2023, learned that the earthquakes significantly impacted a close family member or close friend, or who were exposed to aversive details of the earthquake as part of their job.
* Scoring greater than 47 on the Post-Traumatic Stress Disorder Check List for PTSD symptoms

Exclusion Criteria:

* Acute medical conditions
* Imminent suicide risk
* Expressed acute needs/protection risks
* Indications of severe mental disorders (e.g., psychotic disorders) or cognitive impairment (e.g., severe intellectual disability)
* Severe cognitive impairment (e.g., severe intellectual disability or dementia)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2024-02-25 (Actual); Primary Completion 2025-01-21 (Actual); Study Completion 2025-02-06 (Actual)

PRIMARY OUTCOMES:
Change of the Posttraumatic Stress Disorder Checklist for Diagnostic and Statistical Manual-5 (DSM-5) (PCL-5) over time | change from baseline (one week before the first session of CPT) to post assessment (one week after the last session of CPT); which is expected to last an average of 7 weeks to and 1 months after the intervention
  The PCL-5 is a 20-item questionnaire that assesses the symptoms of PTSD. Items are scored from 0 (not at all) to 4 (extremely) providing a range between 0 and 16. Higher scores indicate higher levels of PTSD symptoms.

SECONDARY OUTCOMES:
Change of the Generalized Anxiety Disorder-7 (GAD-7) over time | change from baseline (one week before the first session of CPT) to post assessment (one week after the last session of CPT); which is expected to last an average of 7 weeks to and 1 months after the intervention
  GAD-7 is a 7-item measure of general anxiety symptoms that measures anxiety symptoms. Each item is scored from 0 (not at all) to 3 (nearly every day) providing a range between 0 and 21. Higher scores indicate higher levels of anxiety.
Change of the World Health Organization (WHO) Well-Being Scale over time | change from baseline (one week before the first session of CPT) to post assessment (one week after the last session of CPT); which is expected to last an average of 7 weeks to and 1 months after the intervention
  WHO Well-being is a 5-item scale that assesses well-being over the last two weeks . Each item is scored from 0 (at no the time) to 5 (all the time) and ranges between 0 and 100 with lower scores indicating worse well-being.
Change of the Patient Health Questionnaire-9 (PHQ-9) over time | change from baseline (one week before the first session of CPT) to post assessment (one week after the last session of CPT); which is expected to last an average of 7 weeks to and 1 months after the intervention
  PHQ-9 is a 9-item questionnaire that aims to measure the depressive symptoms. Each item is scored from 0 (not at all) to 3 (nearly every day) providing a range between 0 and 27. Higher scores indicate more severe depressive symptoms.
Change of the Kessler Psychological Distress Scale (K-10) over time | change from baseline (one week before the first session of CPT) to post assessment (one week after the last session of CPT); which is expected to last an average of 7 weeks to and 1 months after the intervention
  K-10 is a 10-item scale that assesses the psychological distress. Each item is scored from 1 (none of the time) to 5 (all of the time) and ranges between 10 and 50. Higher scores indicate more severe psychological distress.

CONTACTS AND LOCATIONS:
Overall Officials: Büşra Acar, PhD Student, Study Chair — Koç University
Locations (1):
- Koc University, Sarıyer, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moring JC, Dondanville KA, Fina BA, Hassija C, Chard K, Monson C, LoSavio ST, Wells SY, Morland LA, Kaysen D, Galovski TE, Resick PA. Cognitive Processing Therapy for Posttraumatic Stress Disorder via Telehealth: Practical Considerations During the COVID-19 Pandemic. J Trauma Stress. 2020 Aug;33(4):371-379. doi: 10.1002/jts.22544. Epub 2020 Jun 11. PMID 32400911
- [Background] Asmundson GJG, Thorisdottir AS, Roden-Foreman JW, Baird SO, Witcraft SM, Stein AT, Smits JAJ, Powers MB. A meta-analytic review of cognitive processing therapy for adults with posttraumatic stress disorder. Cogn Behav Ther. 2019 Jan;48(1):1-14. doi: 10.1080/16506073.2018.1522371. Epub 2018 Oct 18. PMID 30332919
- [Background] Brown WJ, Dewey D, Bunnell BE, Boyd SJ, Wilkerson AK, Mitchell MA, Bruce SE. A Critical Review of Negative Affect and the Application of CBT for PTSD. Trauma Violence Abuse. 2018 Apr;19(2):176-194. doi: 10.1177/1524838016650188. Epub 2016 Jun 14. PMID 27301345
- [Background] Thomas N, McDonald C, de Boer K, Brand RM, Nedeljkovic M, Seabrook L. Review of the current empirical literature on using videoconferencing to deliver individual psychotherapies to adults with mental health problems. Psychol Psychother. 2021 Sep;94(3):854-883. doi: 10.1111/papt.12332. Epub 2021 Feb 23. PMID 33620133
- See also: General information about CPT — https://www.ptsd.va.gov/professional/treat/txessentials/cpt_for_ptsd_pro.asp